CLINICAL TRIAL: NCT05481346
Title: Psycho-physiological Effects of Multidomain Training in Adults and Older Adults
Brief Title: Effects of Multidomain Training of Health With Aging (Train-Old)
Acronym: Train-Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Pablo Jorge Marcos Pardo, Principal investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UALBIO2022/011
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Sarcopenia; Memory Loss; Muscular Atrophy; Cardiovascular Diseases; Frailty
Keywords: older adults; Healthy aging; Resistance training; cognitive training; cardiovascular training
MeSH Terms: conditions — Sarcopenia; Memory Disorders; Muscular Atrophy; Cardiovascular Diseases; Frailty

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an experimental group that will perform the physical exercise program and a control group that will perform nothing and continue with their normal lifestyle routines, without any physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidomain training group (Experimental): Participants will use free weights and functional materials to work the main muscle groups. In addition, they will perform cardiorespiratory training and cognitive training with proposed tasks. Participants will follow the planned training progression. The researchers will record the number of sets completed and the load lifted for each exercise for each participant and the perception of effort in each class.
  Interventions: Procedure: Multidomain training
- Control group (No Intervention): The control group did not receive a training program and were asked not to modify their physical activity habits.

INTERVENTIONS:
Procedure: Multidomain training — The training program has a duration of 18 weeks with 2 training sessions per week. The training will have a gradual progression of intensity. One day they train two blocks of strength and one block of cognitive exercises and on the second day, they train one block of power, one block of strength+cognitive and one block of aerobic training.
  All sessions are 60 minutes long (10 minutes of warm-up, 40 minutes of training and 10 minutes of cool-down). Classes are in small groups of no more than 8 members.
  Arms: Multidomain training group

SUMMARY:
The current study aims to determine the effect of a multidomain intervention (physical fitness, motivational and cognitive training) on body composition, sarcopenia, cardiovascular health, physical fitness, functional capacity, quality of life, frailty, emotional state and cognitive status in elderly participants, through a randomized controlled trial, to determine its suitability and recommend it as a preventive and health strategy for community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written and dated informed consent to participate in the study.
2. Subject is a male or female between 55 and 90 years of age, inclusive.
3. Subject is in good health as determined by a health history questionnaire and has been provided clearance from their personal physician.
4. Subject is untrained in resistance and aerobic exercise (does not participate in structured physical activity, including walking, more than 3 times per week).
5. Ability to walk independently without any gait aid

Exclusion Criteria:

1. Perform high-intensity aerobic exercise on a consistent basis (>180 min-week).
2. Be performing some other regular and systematic strength training program during the intervention in the first half of 2022.
3. Have a body mass index greater than 35.
4. Have a diagnosis of ischemic heart disease.
5. Have a diagnosis of severe aortic stenosis, uncontrolled arrhythmias, decompensated heart failure or acute myocarditis.
6. Possess uncontrolled blood pressure (TAS >180 and TAD >110).
7. Stroke.
8. Severe peripheral arterial disease.
9. Other illnesses such as recent thromboembolic disease, aortic aneurysm, clinically significant renal or hepatic insufficiency, severe COPD, clinically significant acute infections, severe psychiatric illness, uncontrolled metabolic disease, limiting locomotor pathology or musculoskeletal disease worsened by exercise, hormone therapy at the time or one year prior, being a woman with surgical menopause.
10. Other pathologies that contraindicate the practice of physical exercise, collected in the previous medical examination that all participants must undergo.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-09-18 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Body Weight in Kilograms | Change from Baseline body weight (kg) at 18 weeks
  was measured after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA or InBody equipment to the nearest 0.1 kg.
Height in Meters | Change from Baseline standing height (cm) at 18 weeks
  Standing height without shoes was measured using a Seca 202 stadiometer (Seca, Hamburg, Germany) to the nearest 0.1 cm.
Body Mass Index (BMI) | Change from Baseline Body Mass Index (BMI): (kg/m^2) at 18 weeks
  was calculated as the ratio of weight to squared height in kg/m^2
% Fat Mass | Change from Baseline bioelectrical impedance % fat mass at 18 weeks
  % fat mass was measured after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA or InBody equipment to the nearest 0.1 kg.
Muscle quality sarcopenia | Change from Baseline to 18 weeks
  Sarcopenia will be assessed taking into account the reference values established for muscle quality. The muscle quality will be measure by hand grip strength test. This test will be performance with manual dynamometry (TKK 5401; Scientific Instruments Co., Ltd., Tokyo, Japan). Maximal isometric upper limb strength will be performance by maximal isometric strength. Upper strength will be register by kilogrammes. Higher value show high strength.

SECONDARY OUTCOMES:
Change Blood pressure | Change from Baseline to 18 weeks
  Blood pressure and heart rate will be assessed by means of an automatic device (Colin BP 880, Inc., Tampa, FL). This is noninvasive technique. The result will be register in millimeters of mercury (bood pressure) and number of pulse per minutes (heart rate).
Change Chair stand test | Change from Baseline to 18 weeks
  Chair stand test measure the functional capacity. This is a easy physical test. This test measures the functionality of getting up and sitting down from a chair five times. The participant have to performance the test as faster as possible. The total time is recorded in seconds. A better time indicates better functional ability.
Change Upper and Lower strength | Change from Baseline to 18 weeks
  Maximal isometric upper limb strength will be performance by maximal isometric strength of knee extension and biceps flexion with load cell. Maximal isometric lower limb will be registered in newton. Higher value show high strength.
Health-related quality | Change from Baseline to 18 weeks
  SF-36 quality of life questionnaire
Cardiorrespiratory 6 minutes walk test | Change from Baseline to 18 weeks
  cardiorespiratory endurance test that evaluates the distance covered in 6 minutes.
Change heart rate | Change from Baseline to 18 weeks
  Heart rate will be assessed by means of an automatic device (Colin BP 880, Inc., Tampa, FL). This is noninvasive technique. The result will be register in number of pulse per minutes (heart rate).
Gait speed | Change from Baseline to 18 weeks
  Gait speed will be measure by 4. 6 and 10 meter test. This is easy physical test in with the participant have to walk 4. 6 and 10 metres as faster as possible. The result will be register in seconds. Less time indicates better functional ability.
Time up and go test change | Change from Baseline to 18 weeks
  Time up and go test measure the functional capacity of getting up, walking and sitting down form a chair. Participant have to performance this test as faster as possible. This is a easy physical test. Total seconds are records. Less seconds indicates better functional ability.
Short physical performance battery (SPPB) | Change from Baseline to 18 weeks
  Short physical performance battery (SPBB) include three test (balance, chair stand test and gait speed) and report a final score. Chair stand test and gait speed were describe in other outcome. Balance test is a easy physical test. The participant must maintain three balancing positions for 10 seconds to overcome it. Each test offers a different score. Higher score show better functional capacity.
Fragility | Change from Baseline to 18 weeks
  Frailty will be defined in relation to Fried's frailty phenotype (Fried et al., 2001), based on 5 criteria: unintentional weight loss, exhaustion, weakness, slow walking speed and low physical activity.
Satisfaction with life | Change from Baseline to 18 weeks
  The Satisfaction with Life Scale is a 4-item instrument with a Likert-type scale ranging from 1 to 7 points measuring overall subjective happiness by means of statements in which participants rate themselves or compare themselves with others. Two items ask people to describe themselves using absolute rating criteria of their lives or rating criteria with respect to others, while the other two items present brief descriptions of happy or unhappy people and respondents are asked to indicate the degree to which they identify with that description.
Depression | Change from Baseline to 18 weeks
  Depression will be measured through the Center for Epidemiological Studies Depression Scale-Revised (CESD-R) (Van Dam & Earleywine, 2011), is a 20-item questionnaire that can be used to measure levels of depressive symptoms among elderly participants. The CESD-R consists of 16 items of negative affect and 4 items of positive affect.
Cognitive flexibility | Change from Baseline to 18 weeks
  the Stroop test measures the ability to classify information selectively. It consists of 3 phases and requires discerning between colors and words without making mistakes.
Attention test | Change from Baseline to 18 weeks
  the Trail Making test will also assess flexibility of thought and visuospatial ability. It consists of joining numbers and words in a numerical sequence without error.
PSQ test | Change from Baseline to 18 weeks
  To evaluate the factors that influence the general state of health, specifically stress. It evaluates six factors: Tension-Instability-Fatigue; Social Acceptance of Conflict; Energy and Fun; Overload; Satisfaction for self-fulfillment; Fear and anxiety.
TMMS-24 | Change from Baseline to 18 weeks
  Trait-Meta Mood Scale (TMMS) emotional states

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Jorge Marcos Pardo, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Pablo Jorge Marcos Pardo, Almería, Spain

IPD SHARING:
Plan to Share IPD: No
Once the data are published, the data can be requested and will be made available to other researchers.